CLINICAL TRIAL: NCT02158325
Title: Appropriate Capsulorhexis Size Results in Better Capsular Outcome When Treating Pediatric Cataract: A Randomized Controlled Trial
Brief Title: Capsulorhexis Size and Capsular Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Ophthalmologist, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2010-China6
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Congenital Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3.0-3.9 mm (Active Comparator): pediatric cataract surgery performed with different anterior capsulorhexis sizes (3.0-3.9 mm in diameter)
  Interventions: Procedure: anterior capsulorhexis sizes
- 4.0-5.0 mm (Experimental): pediatric cataract surgery performed with different anterior capsulorhexis sizes (4.0-5.0 mm in diameter)
  Interventions: Procedure: anterior capsulorhexis sizes
- 5.1-6.0 mm (Active Comparator): pediatric cataract surgery performed with different anterior capsulorhexis sizes (5.1-6.0 mm in diameter)
  Interventions: Procedure: anterior capsulorhexis sizes

INTERVENTIONS:
Procedure: anterior capsulorhexis sizes — Pediatric cataract surgery performed with different anterior capsulorhexis sizes (3.0~3.9, 4.0~5.0, 5.1~6.0 mm in diameter)

SUMMARY:
Different capsulorhexis size results in different capsular outcome when treating pediatric cataract, and there should be an appropriate capsulorhexis size for the best capsular outcome.

DETAILED DESCRIPTION:
Numerous studies have reported that ideal anterior capsulorhexis size is 4.5-5.0 mm with the capsulorhexis edges covering IOL optic surface because it can inhibit the proliferation and migration of remnant lens epithelial cells (LEC). But there are no reports investigating the relationship between the capsulorhexis size and the capsular outcome after pediatric cataract surgery. Therefore, the aim of the current study is to prospective evaluate the capsular outcomes of three controlled groups receiving different anterior capsulorhexis sizes (3.0-3.9, 4.0-5.0, 5.1-6.0 mm in diameter).

ELIGIBILITY:
Inclusion Criteria:

* Age< 2 years
* performed cataract surgery without IOL implantation
* without capsular fibrosis, glaucoma, ocular trauma, corneal disorders before surgery
* No other corneal and systemic abnormalities
* Written informed consents provided

Exclusion Criteria:

* Patients with glaucoma, ocular trauma, corneal disorders, persistent hyperplastic primary vitreous, rubella, Lowe syndrome, capsular fibrosis
* Cases with surgical complications
* those who can't dilute pupil normally postoperation or can't complete the follow-up

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Mean area of anterior/posterior capsulorhexis opening | two years

SECONDARY OUTCOMES:
the ratio of opacity accounting for posterior capsulorhexis opening at different visits | two years
The area change of anterior/posterior capsulorhexis opening | two years

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Luo L, Lin H, Chen W, Wang C, Zhang X, Tang X, Liu J, Congdon N, Chen J, Lin Z, Liu Y. In-the-bag intraocular lens placement via secondary capsulorhexis with radiofrequency diathermy in pediatric aphakic eyes. PLoS One. 2013 Apr 24;8(4):e62381. doi: 10.1371/journal.pone.0062381. Print 2013. PMID 23638058
- [Background] Lin H, Chen W, Luo L, Zhang X, Chen J, Lin Z, Qu B, Zhan J, Zheng D, Zhong X, Tian Z, Liu Y; Study Group of CCPMOH. Ocular hypertension after pediatric cataract surgery: baseline characteristics and first-year report. PLoS One. 2013 Jul 29;8(7):e69867. doi: 10.1371/journal.pone.0069867. Print 2013. PMID 23922832
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- See also: Homepage of Zhongshan Ophthalmic Center — http://www.gzzoc.com/